CLINICAL TRIAL: NCT04595292
Title: Validity Reliability of The Dubousset Functional Test in Older Adults
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ayşe Abit Kocaman, Principal Investigator, Kırıkkale University
Other Study IDs: The Dubousset Functional Test
Record Dates: First submitted 2020-10-09; First posted 2020-10-20 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Aging; Fall; Balance; Distorted
MeSH Terms: interventions — Aging; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- older adults, assessment
  Interventions: Other: older adults, assessment

INTERVENTIONS:
Other: older adults, assessment — Dubousset Function Test, 3-m backwards walk test, timed up and go test,Tinnetti Balance and Gait Test, Berg BalanceTest, Functional Reach Test

SUMMARY:
Postural deformity and postural instability that occur with aging are risk factors for falling.

In the literature, there are many scales that evaluate balance and functional performance in older adults. However there is no validity and reliability study of Dubousset Function Test developed to evaluate balance and functional performance of older adults. For this reason, the aim of study is to examine the validity and reliability of Dubousset Function Test in older adults.

DETAILED DESCRIPTION:
However, postural deformity and postural instability that occur with aging are risk factors for falling. In studies examining the relationship between postural instability and spinal curvatures, it was stated that the balance and functional performance of patients with increased kyphosis were affected. Increased thoracic kyphosis and lumbar lordosis loss in geriatric individuals, degenerative spinal deformities are common and functional limitations lead to negative clinical consequences such as an increase in the risk of falls or fractures and impaired quality of life.

Dubousset Functional Test (DFT); A conceptually practical four-component assessment test has been proposed by Dr. Jean Dubousset to assess the functional capacity of adult individuals. The validity of the test was made in individuals with spinal deformity. DFT; It consists of four components: getting up from a chair without arms and walking 5 meters forward and backward, descending and climbing steps, transition from standing to sitting on the ground, and the dual task test in which the individual walks while counting down from 50 at the same time.

In the literature, there are many scales that evaluate balance and functional performance in elderly individuals.However, there is no validity and reliability study of Dubousset Function Test developed to evaluate balance and functional performance of adult individuals in elderly individuals. For this reason, the aim of study is to examine the validity and reliability of Dubousset Function Test in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over,
* Volunteering to participate in research
* No cooperation and communication problem

Exclusion Criteria:

* Individuals with neurological and orthopedic problems
* Uncontrollable hypertension
* Those with cardiac disease
* Those with cooperation and communication problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Individuals aged 65 and over, Volunteering to participate in research, No cooperation and communication problem
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Dubousset Function Test | first day
  The four components of the DFT included (1) the Up Walking Test: participants rose without assistance from a and seated position in a chair that did not have arms, walked 5 meters (500 cm) forward before stopping, walked backwards 5 meters, and sat again without assistance; (2) the Steps Test: from a starting position 50 cm away, volunteers climbed three stairs, turned around on the third step (top), and walked down the three steps; (3) Down and Sitting Test: from a standing position, participants sat on the ground and stood up again, using assistance as needed; (4) Dual-Tasking Test: participants walked 5 meters forward, turned around, and walked 5 meters back to the starting position while performing a working memory test (counting down from 50 by intervals of 2).
timed up and go test | first day
  A standard chair is used for testing. First, the patient is asked to sit on the chair. The patient is then asked to stand up and walk regularly at a distance of 3 meters with a predetermined length, then return to the chair after 3 meters.
3-m backwards walk test, | first day
  A distance of 3 m is measured and marked with black tape. Individuals are asked to follow the heel and black band.
  With the 'start' command they are asked to walk backwards quickly. When the distance of 3 m is completed, a stop is instructed. Individuals are not allowed to run during the test. They are allowed to look back if they wish. The assessor walks behind individuals throughout the test. The test is repeated 3 times, the averages are recorded
Tinetti Balance and Gait Test | first day
  In the test used to evaluate balance, walking score is maximum 12 points, balance score is maximum 16 points and a total of 28 points.
Berg Balance Test | first day
  The BBS consists of 14 items to directly monitor the maintenance of body balance during performance
Funtional Reach Test | first day
  It is used to measure both the balance of the individual functionally and the amount of dynamic reach

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diebo BG, Challier V, Shah NV, Kim D, Murray DP, Kelly JJ, Lafage R, Paulino CB, Passias PG, Schwab FJ, Lafage V. The Dubousset Functional Test is a Novel Assessment of Physical Function and Balance. Clin Orthop Relat Res. 2019 Oct;477(10):2307-2315. doi: 10.1097/CORR.0000000000000820. PMID 31135543